CLINICAL TRIAL: NCT05754424
Title: A Phase 1, Single Centre, Single Dose, Randomised, Double-blind, Two-way Crossover, Glucose Clamp Study Investigating the Pharmacodynamics, Pharmacokinetics, and Safety of Ultra-rapid-acting Concentrated Insulin Aspart AT278 in Comparison to Standard Insulin Aspart NovoRapid® With an Additional Open Comparison to Humulin® R U-500 in Participants With Type 2 Diabetes.
Brief Title: AT278, NovoRapid® and Humulin® R (U500) in Glucose Clamp Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arecor Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARE-278-104; 2022-001984-28 (EudraCT Number)
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT278 (Experimental): Single subcutaneous injection of 0.5 U/kg
  Interventions: Drug: AT278; Drug: NovoRapid; Drug: Humulin R 500 UNT/ML Injectable Solution
- NovoRapid (Active Comparator): Single subcutaneous injection of 0.5 U/kg
  Interventions: Drug: AT278; Drug: NovoRapid; Drug: Humulin R 500 UNT/ML Injectable Solution

INTERVENTIONS:
Drug: AT278 — Concentrated rapid acting insulin aspart
Drug: NovoRapid — Rapid-acting insulin aspart
Drug: Humulin R 500 UNT/ML Injectable Solution — Regular human insulin

SUMMARY:
This is a phase 1, single dose, randomised, double-blind, two-way crossover study to compare ultra-rapid-acting concentrated insulin aspart AT278 (U500/mL) with standard insulin aspart NovoRapid® (U100/mL) in participants with T2D. Participants and Investigators will be blinded to both study interventions. Humulin® R U-500 (U500/mL), a highly concentrated regular human insulin, will be used as an open-label comparator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for at least 180 days prior to the day of screening
* Haemoglobin A1C (HbA1c) concentration of ≤9.5% (≤80 mmol/mol) at screening.
* BMI within the range of 25 - 45 kg/m2 (both inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs or related products
* Clinically significant concomitant disease or abnormal lab values
* Severe asthma or chronic obstructive pulmonary disease (GOLD III and IV), or lower if requiring high dose of corticosteroids or beta2-adrenergic agonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate-time curve of insulin aspart | 0 to 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Unit, Medical University of Graz, Graz, Austria